CLINICAL TRIAL: NCT05653219
Title: A Phase 3 Randomized, Double-blind Study of Ianalumab (VAY736) Versus Placebo in Addition to Eltrombopag in Patients With Primary Immune Thrombocytopenia (ITP) Who Had an Insufficient Response or Relapsed After First Line Steroid Treatment (VAYHIT2)
Brief Title: A Study of Efficacy and Safety of Ianalumab Versus Placebo in Addition to Eltrombopag in Primary Immune Thrombocytopenia Patients Who Failed Steroids
Acronym: VAYHIT2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736Q12301; 2024-512890-28-00 (Other: EU CTIS)
Record Dates: First submitted 2022-11-23; First posted 2022-12-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Primary immune thrombocytopenia (ITP),; ianalumab; VAY736; B-cell depletion; B-cell Activating Factor Receptor (BAFF-R) blockade; eltrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — ianalumab; eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment arm 1 (Experimental): Participants will receive eltrombopag and ianalumab lower dose
  Interventions: Biological: Ianalumab; Drug: Eltrombopag
- Treatment arm 2 (Experimental): Participants will receive eltrombopag and ianalumab higher dose
  Interventions: Biological: Ianalumab; Drug: Eltrombopag
- Treatment arm 3 (Placebo Comparator): Participants will receive eltrombopag and placebo
  Interventions: Drug: Eltrombopag; Drug: Placebo

INTERVENTIONS:
Biological: Ianalumab — Concentrate for solution for infusion for intravenous use
  Other Names: VAY736
  Arms: Treatment arm 1; Treatment arm 2
Drug: Eltrombopag — Film-coated tablet for oral use
  Other Names: ETB115
Drug: Placebo — Concentrate for solution for infusion for intravenous use.
  Arms: Treatment arm 3

SUMMARY:
The purpose of this study is to evaluate the effect of two different doses of ianalumab added to eltrombopag to prolong Time to Treatment Failure (TTF) in adults with primary ITP who failed previous first-line treatment with steroids.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded phase 3 study to assess efficacy and safety of two different doses of ianalumab versus placebo in addition to eltrombopag in adults with primary ITP (platelet count <30 G/L) who failed previous first-line treatment with corticosteroids.

After completion of the screening period, the participants will enter the randomized treatment period (ianalumab/placebo with eltrombopag) followed by the eltrombopag tapering period. Afterwards, all participants will enter the follow-up period to be monitored for efficacy and safety or safety only depending on how the participants responded to the study treatment.

ELIGIBILITY:
Key Inclusion criteria

1. Male or female patients aged 18 years and older on the day of signing the informed consent.
2. A signed informed consent must be obtained prior to participation in the study.
3. A diagnosis of primary ITP, with insufficient response to, or relapse after a first-line corticosteroid therapy ± IVIG.
4. Patient with platelet count <30G/L (whom eltrombopag is clinically indicated as per physician's discretion) and with no contraindication to receive eltrombopag

Key Exclusion criteria

1. ITP patients who received second-line ITP treatments (other than steroid therapy± IVIG) including splenectomy. However, patients exposed to thrombopoietin receptor agonists (TPO-RAs) for a limited time (max one week) before screening are eligible.
2. Patients with key lab abnormalities and patients with Evans syndrome or any other cytopenia, (patients with low grade anemia related to bleeding or iron deficiency are eligible).
3. Patients with history of clinically significant hematological disorders, or with marked altered hematologic parameters
4. Patients with current or history of life-threatening bleeding
5. Patient that are Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV), Hepatitis B surface Antigen (HBsAg)/ Hepatitis B core antibody (HBcAb)-positive. HBcAb-positive patients can be enrolled if HBsAg negative, HBV DNA negative, no pre-existing liver fibrosis is present and antiviral prophylaxis is given
6. Patients with known active or uncontrolled infection requiring systemic treatment during screening period
7. Patients with hepatic impairment
8. Patients with concurrent coagulation disorders and/or receiving antiplatelet or anticoagulant medication with an exemption of low dose of acetylsalicylic acid (≤150 mg daily)
9. Nursing (breast feeding) or pregnant women

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
Time from randomization until treatment failure | Randomization to until end of study (up to 39 months after randomization of last participant)
  Time from randomization until treatment failure is defined as the time from randomization date until the first of the following events indicative of treatment failure:
  * platelet count below 30 G/L
  * start of a new ITP treatment
  * need for a rescue treatment
  * ineligibility to taper or inability to discontinue eltrombopag
  * death

SECONDARY OUTCOMES:
Stable response at 6 months (Key Secondary Endpoint) | At 6 months
  Percentage of participants with at least 3 platelet count collected at month 6 (between study days 121 and 183 and at least 75% of platelet counts qualified as a response).
Complete Response rate at each timepoint | Randomization to until end of study (up to 39 months after randomization of last participant)
  Percentage of participants with any platelet count of at least 100 G/L in the absence of rescue treatment or new ITP treatment
Response rate at each timepoint | Randomization to until end of study (up to 39 months after randomization of last participant)
  Percentage of participants with any platelet count of at least 50 G/L in the absence of rescue treatment or new ITP treatment
Best response rate across all timepoints | Randomization to until end of study (up to 39 months after randomization of last participant)
  Percentage of participants with a best response rate of either response or complete response
Time to first response/time to first complete response | Time from randomization up to the longest observed treatment period duration
  Time from randomization to date of first response and time from randomization to date of first complete response
Duration of response | Randomization to until end of study (up to 39 months after randomization of last participant)
  Time from achievement of response to treatment failure.
Stable response at 1 year | At 1 year
  Percentage of participants with at least 2 platelet count collected at year 1 (between study days 296 and 379 and at least 66% of platelet counts qualified as a response).
Duration of complete response | Randomization to end of study (up to 39 months after randomization of last participant)
  Time from achievement of complete response to loss of complete response stable response at 1 year period
Rate of participants who successfully taper and discontinue eltrombopag in each treatment arm | up to week 24
  Probability to be treatment failure-free (as defined for the primary efficacy endpoint)
Percentage of participants with bleeding events according to World Health Organization (WHO) | Randomization to until end of study (up to 39 months after randomization of last participant)
  Percentage of participants reporting bleeding events according to WHO bleeding scale
Number of participants receiving rescue treatment | Randomization to until end of study (up to 39 months after randomization of last participant)
  Number of participants who are in need of rescue treatment in each treatment arm
Percentage of participants receiving rescue treatment | Randomization to until end of study (up to 39 months after randomization of last participant)
  Percentage of participants who are in need of rescue treatment
Change from baseline in the frequency of CD19+ B-cell counts | Randomization to until end of study (up to 39 months after randomization of last participant)
  Post-baseline frequency of CD19+ B-cell counts (percentage within CD45) compared to baseline
Change from baseline in the absolute number of CD19+ B-cell counts | Randomization to until end of study (up to 39 months after randomization of last participant)
  Post-baseline absolute number of CD19+ B-cell counts compared to baseline
Change from baseline on T-score of the PROMIS SF v1.0 Fatigue 13a | From screening (baseline) until end of study (up 39 months after randomization of last participant)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Fatigue 13a includes 13 items that assess fatigue in adults.
Change from baseline in ITP PAQ domain scores of symptoms, fatigue, bother (uncomfortable), activity | From screening (baseline) until end of study (up 39 months after randomization of last participant)
  The ITP-PAQ is a 44 item scale for measuring HRQoL in adults with ITP across ten scales: Symptoms, Bother-Physical Health, Fatigue/Sleep, Activity, Fear, Psychological Health, Work, Social Activity, Women´s Reproductive Health, overall QoL. Each item is rated on a Likert type scale. Each scale is scored from 0 to 100. Higher scores represent better HRQoL.
Time to first occurence of B-cell recovery defined as ≥80% of baseline ≥50 cells/µL | Randomization to until end of study (up to 39 months after randomization of last participant)
  Time to B-cell recovery defined as ≥80% of baseline or ≥50 cells/µL
Change from baseline in immunoglobulins | Randomization to until end of study (up to 39 months after randomization of last participant)
  Change from baseline in immunoglobulin levels
PK parameters: AUClast | After first dose (pre-dose, EOI, 168, 336 and 504 hours post dose) and after last dose (pre-dose, EOI, 336, 672, 2016, 3360 hours post dose)
  AUClast: Area under the curve from time zero to the last measurable concentration sampling time (tlast)
PK parameters: AUCtau | After first dose (pre-dose, EOI, 168, 336 and 504 hours post dose) and after last dose (pre-dose, EOI, 336, 672, 2016, 3360 hours post dose)
  AUCtau: Area under the curve calculated to the end of a dosing interval (tau)
PK parameters: Cmax | After first dose (pre-dose, EOI, 168, 336 and 504 hours post dose) and after last dose (pre-dose, EOI, 336, 672, 2016, 3360 hours post dose)
  Maximum (peak) observed plasma, blood, serum or other body fluid drug concentration
PK parameters: Tmax | After first dose (pre-dose, EOI, 168, 336 and 504 hours post dose) and after last dose (pre-dose, EOI, 336, 672, 2016, 3360 hours post dose)
  Time to reach maximum (peak) observed plasma, blood, serum or other body fluid drug concentration
PK parameters: Accumulation ratio Racc | After last dose (pre-dose, EOI, 336, 672, 2016, 3360 hours post dose)
  Accumulation ratio calculated using AUC values obtained after the last and first dose
Incidence of anti-ianalumab antibodies in serum (ADA assay) over time | up to week 33
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants assessing the immunogenicity of ianalumab
Titer of anti-ianalumab antibodies in serum (ADA assay) over time | up to week 33
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants assessing the immunogenicity of ianalumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (70):
- United States (9):
  - Yuma Regional Medical Center, Yuma, Arizona
  - University of Colorado Anschutz, Aurora, Colorado
  - NorthShore University Health System, Evanston, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Hematology Oncology Association of Rockland, Nyack, New York
  - Montefiore Medical Center, The Bronx, New York
- Novartis Investigative Site, CABA, Argentina
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Yvoir, Namur
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
- China (7):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Binzhou, Shandong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Tianjin
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- France (2):
  - Novartis Investigative Site, Blois
  - Novartis Investigative Site, Le Mans
- Germany (4):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Dresden
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- India (2):
  - Novartis Investigative Site, Rishikesh, Uttarakhand
  - Novartis Investigative Site, Kolkata, West Bengal
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Trieste, TS
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kofu, Yamanashi
  - Novartis Investigative Site, Kumamoto
- Malaysia (6):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Subang Jaya, Selangor
  - Novartis Investigative Site, George Town
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Kuala Selangor
- Mexico (3):
  - Novartis Investigative Site, Saltillo, Coahuila
  - Novartis Investigative Site, Morelia, Michoacán
  - Novartis Investigative Site, Monterrey, Nuevo León
- Netherlands (2):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Utrecht
- Philippines (2):
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Quezon
- Romania (2):
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Timișoara
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Jeollanam
  - Novartis Investigative Site, Seoul
- Spain (2):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Salamanca
- Novartis Investigative Site, Taoyuan District, Taiwan
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Ankara, Bilkent Cankaya
  - Novartis Investigative Site, Aydin, Efeler
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Izmir
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Cuker A, Stauch T, Cooper N, Al-Samkari H, Michel M, Ghanima W, Urban P, Fronczek J, Foster M, Weill M, Zhang L, Hou M, Zander T, Sharif A, Sun J, Nath UK, Schutgens R, Rossi E, Deleu L, Cervinek L, Yoon JH, Chang H, Ruchutrakool T, Iino M, Goto T, Zaja F; VAYHIT2 Investigators. Ianalumab plus Eltrombopag in Immune Thrombocytopenia. N Engl J Med. 2025 Dec 9. doi: 10.1056/NEJMoa2515168. Online ahead of print. PMID 41363800